CLINICAL TRIAL: NCT04957420
Title: Neupro's Multicenter and Prospective Observation of Safety and Efficacy in Chinese Mainland Idiopathic Parkinson's Disease in Real World Practice
Brief Title: The Practical Effect of Neupro
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: D2021060
Record Dates: First submitted 2021-06-27; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neupro gruop: Patients using Neupro according to the standard clinical practice of therapists
  Interventions: Drug: Neupro

INTERVENTIONS:
Drug: Neupro — Rotigotine Patches

SUMMARY:
This is a multicenter, prospective, non intervention post marketing surveillance study conducted in Chinese mainland. The main objective was to evaluate the safety characteristics of rotigotine patch in the treatment of Chinese adult patients with idiopathic Parkinson's disease in real world clinical practice.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a long-term, chronic, progressive and disabling disease, which affects millions of patients worldwide. The incidence rate of Parkinson's disease is about 20/100000 per year. With the increase of age (65 years old and above), the incidence rate of the population increased significantly, reaching >100/100000 per year . The average age of onset is 58 to 62 years old, and the prevalence rate of people over 50 years old is about 1%. Similar to the incidence rate, the prevalence of Parkinson's disease increases with age. It is 1.4% at 55 years old, and 4.3% in 85 years old and above.

The main clinical symptoms of Parkinson's disease include tremor, myotonia, motor retardation, postural reflex disorders and gait disorders, as well as a variety of other motor, mental, sensory and autonomic neuropathy. Depressive symptoms of Parkinson's disease are very common in patients. In the progressive stage of the disease, patients may have dementia symptoms. Autonomic nervous system involvement may cause orthostatic hypotension, paroxysmal flushing, thermoregulation disorders, constipation, dysphagia, bladder and sexual dysfunction. Involvement of dopaminergic pathways in the thalamus and spinal cord may lead to sensory abnormalities.

The etiology of Parkinson's disease remains unclear. However, it is generally considered to be a progressive degenerative disease, which gradually erodes the brain stem, basal ganglia structure and its projection system. Pathological studies have found that there are loss of dopaminergic neurons in substantia nigra and neurons in locus coeruleus and raphe nucleus, deposition of Lewy bodies and activation of glial cells. Basic studies suggest that oxidative damage of specific neurons in basal ganglia is one of the potential causes of idiopathic Parkinson's disease, and aging and genetic factors are also the main causes of the disease

Predisposing factors.

Rotigotine ((6S) - 6 - {propyl [2 - (2-thienyl) ethyl] amino} - 5,6,7,8-tetrahydro-1-naphthol) is the left-handed enantiomer of chiral aminotetrahydronaphthalene compounds. Rotigotine is a dopamine receptor agonist. Its dosage form is designed as a transdermal drug delivery system, which can continuously release rotigotine within 24 hours. Transdermal drug delivery system, which continuously releases dopamine receptor agonists (such as rotigotine) in a non-invasive manner. Rotigotine has been approved by global health agencies for the treatment of early and advanced Parkinson's disease. Overall, ushib or authorized partners have market licenses for rotigotine transdermal patches for Parkinson's disease in 70 countries. A detailed description of the preclinical and clinical experience of rotigotine can be found in the investigator's manual.

From February 15, 2006 to February 15, 2020, a total of 7878 participants used rotigotine as part of the clinical development plan. No treatment-related risk was found in the longest 6-year long-term open study. Other safety features of rotigotine, including clinical and post marketing data, can be found in the investigator's manual.

According to the current policy of the Chinese government, multinational pharmaceutical companies operating in China should implement drug safety monitoring within five years after obtaining the registration certificate of imported drugs. This kind of research is called focused drug monitoring (IDM), which aims to investigate the safety and clinical application of products, including expected and unexpected adverse drug reactions (ADRs); Specific adverse reactions / events are related, incidence rate, severity, risk and so on. The incidence of ADR in special groups, including pregnant women, children, the elderly, patients with liver and kidney damage, specific race, patients with specific genetic tendency or specific complications, and other people who lack safety data of pre marketing clinical studies; Other safety problems related to drug use, packaging and quality were observed. During IDM, general population monitoring should be used unless there are other requirements for special reasons (such as requirements or permission of drug regulatory agencies). Observational studies are recommended. According to the data collection method, prospective study is recommended. However, in order to collect data as comprehensively as possible, prospective and retrospective studies can also be combined. Literature research can be used as a brief supplement to key monitoring methods. In order to avoid information collection bias during IDM, case selection should be continuous, such as collecting information of all patients using drugs in a specific time period and fixed medical institutions; Other biases should also be considered in planning. According to the requirements of China's State Food and Drug Administration (CFDA) / State Drug Administration (nmpa), Neupro®（ The safety characteristics of rotigotine patches need to be evaluated using a sample of at least 3000 patients.

The purpose of this non intervention study (NIS) was to evaluate the safety of rotigotine patch in adult patients with idiopathic Parkinson's disease according to the instructions in routine clinical practice, so as to meet the regulatory requirements of Chinese health institutions. This study will collect and monitor all adverse events (AE). Evidence of the efficacy and use of rotigotine patches in the real world will also be collected with AE.

ELIGIBILITY:
Inclusion Criteria:

-

Patients must meet the following selection criteria to enter the non intervention study:

1. The decision of the treatment doctor to prescribe rotigotine patch has nothing to do with whether to participate in the non intervention study.
2. The patient or his legal representative can understand the informed consent of the patient data.
3. The informed consent form of patient data shall be signed and dated by the patient or his legal representative.
4. The patient is over 18 years old.
5. The patient was diagnosed as idiopathic Parkinson's disease

Exclusion Criteria:

-

Patients meeting any of the following criteria should be excluded from the study:

1. For any reason, the researcher (therapist) thinks that the patient is not suitable to participate in this study.
2. Patients had received rotigotine patch for more than 4 weeks before study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient was diagnosed as idiopathic Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
(serious) adverse events (AE) and (serious) adverse drug reactions (ADRs) | in 12 weeks
  (serious) adverse events (AE) and (serious) adverse drug reactions (ADRs)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijin, China

IPD SHARING:
Plan to Share IPD: No